CLINICAL TRIAL: NCT02119767
Title: Study to Detect Biomarker Gradients in Coronary Arteries Using the Liquid Biopsy System
Acronym: CS1
Status: Completed | Type: Observational
Sponsor: PlaqueTec Ltd (Industry)
Collaborators: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: CE002
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Coronary Heart Disease
Keywords: Atherosclerosis
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Natural gradients: Patients requiring an elective PCI who present with either non-ST-segment elevation myocardial infarction (NSTEMI) or chronic stable angina who will have natural gradients sampled using the LBS
- Induced gradients: Patients requiring an elective PCI who present with either non-ST-segment elevation myocardial infarction (NSTEMI) or chronic stable angina who will have induced gradients sampled using the LBS

SUMMARY:
The Liquid Biopsy System (LBS) is a new catheter (thin tube) designed for sampling blood directly from coronary arteries. These arteries supply blood to muscles of the heart and can become blocked by 'plaques' leading to chest pain (angina) and heart attacks. Recent research has shown that development of ' plaques' inside coronary arteries is controlled by chemicals (biomarkers) released into the blood from damaged areas of the artery wall. The LBS is designed to collect blood samples at the exact site of plaque formation. By testing these blood samples for biomarkers of plaque formation, it is hoped that new diagnostic tests and treatments for heart disease may be developed. The proposed investigation is use the LBS in humans to detect these biomarkers. The safety of the LBS has already been demonstrated in both human and animal studies. The study will enroll 70 patients with coronary artery disease who are undergoing routine percutaneous coronary intervention (PCI). PCI is a procedure used to open up a blocked coronary artery. It uses a catheter on the end of which is a special balloon that is inflated inside the blocked artery to open up the vessel and restore blood flow. A small metal spring (stent) is usually inserted to keep the blood vessel open. This study will test if the LBS device, when used just prior to a PCI procedure, can detect biomarkers released by diseased coronary arteries. The study will also determine if the presence of these biomarkers is linked to the long term health of the patient. The study will take place at Papworth Hospital, over a period of approximately 8 months (including telephone based patient followup calls 30 days, 6 months, 1, 2 and 3 years after the procedure to determine patient health).

DETAILED DESCRIPTION:
The purpose of this Clinical Investigation is to use the PlaqueTec Liquid Biopsy System (LBS) to determine which biomarkers detected locally within the coronary artery can give information on the state of atherosclerotic disease. The LBS is a novel CE-marked class III coronary catheter designed for sampling blood directly from the coronary arteries. The LBS is unique in that it can capture "gradients" of biological molecules within the coronary artery and by analysing the samples it collects it can unequivocally identify which biomarkers have been locally released within the coronary artery. The samples can then be analysed for a variety of biomarkers using standard analytical techniques. Cardiologists should find this of great benefit as recent studies have shown that coronary artery disease is controlled and directed by the release of specific biological molecules into the blood from diseased areas of the coronary arteries. The safety and performance of the LBS has been proved previously in a recent First In Man study. The Clinical Investigation study will enroll 70 patients and will be observational in nature. The study is designed to use the device in its intended application (i.e. as an adjunct to a PCI procedure, such as the deployment of a stent) and to collect biomarker gradients released locally within the coronary artery. It will then follow up on the health status of the patients and see if the release of certain biomarkers is associated with particular clinical outcomes. The device will be used to look for locally released biomarkers at two different stages of the deployment of a stent, i.e. before and after its deployment. The first stage is prior to the deployment of the stent and the LBS will collect blood samples to look for the release of "natural" biomarkers gradients, i.e. those biomarkers that are naturally released during the progression and development of diseased regions within the artery. The second stage is to use the LBS to collect blood samples across a diseased artery that has just be perturbed (by "pre-ballooning", a procedure carried out just prior to stent insertion) and will looked for "induced" biomarker gradients, i.e. those molecules that are released by a diseased plaque when it ruptures. The insights gained by collecting biomarker gradients at these two stages will give very important information on what causes a region of artery to become diseased and how diseased portions of the artery affect the blood and cause heart attacks. The samples that are collected by the LBS in the above clinical settings will be analysed for a series of biomarker gradients previously selected by PlaqueTec' s Scientific Advisory Panel (SAP) for their potential role in causing atherosclerosis. The data collected by the LBS will be for research only and will not be used to affect the patient treatment. In summary, the LBS study will deliver completely new insights into coronary artery disease and will significantly increase the understanding of this hugely significant disease. Patients who need an elective percutaneous transluminal interventional coronary procedure will be considered for this study. Patients requiring emergency interventional procedures will be excluded. The study duration is estimated to be about 8 months with a three year follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects that are candidates for percutaneous transluminal interventional coronary procedures
2. Subjects undergoing elective PCI
3. Subjects presenting for PCI after NSTEMI
4. Subjects who have been preloaded with dual antiplatelet therapy (aspirin and clopidogrel (or prasugrel or ticagrelor)) as per usual local PCI practice.
5. Subjects who are willing and able to sign an informed consent.

Exclusion Criteria:

1. Subjects for whom the LBS is contra-indicated:

   1. The LBS is contraindicated for use in severely stenosed, excessively tortuous or calcified coronary vessels.
   2. The LBS is contraindicated in coronary vessels with a reference diameter of less than 2.5 mm.
   3. The LBS is contraindicated for use in regions of coronary vessels that contain a stent.
   4. The LBS is contraindicated for use in the carotid arteries, cerebral vessels or any of their side branches.
   5. The LBS is contraindicated for use with patients in whom anticoagulant or antiplatelet therapy is contraindicated, or have uncorrected bleeding disorders or an allergy to heparin.
   6. Use of the LBS is contraindicated in patients with ongoing sepsis that is considered relevant to cardiac catheterization.
   7. The LBS is contraindicated for use in the acute phase of an ST Segment Elevation Myocardial Infarction, in patients with severe hemodynamic instability or shock.
   8. The LBS is contraindicated for use in the presence of angiographic evidence of intracoronary thrombus.
2. Subjects who are unwilling or unable to sign an informed consent
3. Subjects undergoing immunosuppressive therapies
4. Severe left ventricular dysfunction (left ventricular ejection fraction <30%)
5. Cardiogenic shock
6. PCI target in left main stem
7. PCI target lesion with low pre-procedure chance of success or high pre-procedure risk of complication (e.g. chronic total occlusion, thrombus load)
8. Subjects <18 years (there is no upper age limit but there is a requirement that patients are considered to be "fit" enough by the operating cardiologist for the LBS procedure to not cause significant additional risk)
9. Pregnancy
10. Contraindication to dual antiplatelet therapy or inability to take dual antiplatelet therapy for at least 4 weeks post-procedure
11. Serum creatinine above 125 µmol/L.(i.e. the upper limit for normal)
12. Subjects on warfarin at the time of procedure
13. Subjects with active chronic inflammatory disease, e.g. systemic lupus erythematosus, rheumatoid arthritis, seropositive arthropathies and known seropositivity to HIV, Hepatitis B or Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited at secondary care cardiology facilities. All subjects who need a percutaneous transluminal interventional coronary procedure (excluding those with an ST elevation myocardial infarction) will be considered for this study.
  Potential participants will be identified from pre-admission clinic lists and screened for suitability by members of the clinical team. Eligible patients will be approached for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Local release of biomarkers by diseased regions of the coronary artery | 2 years
  That biomarkers are released locally by diseased regions of the coronary artery (either naturally or during pre-ballooning for stenting) of patients with cardiovascular disease (CVD) and detectable using the LBS and associated assays

SECONDARY OUTCOMES:
Clinical outcome of detected coronary gradients (by telephone for all patients) | 3 years 8 months
  This will test whether the local release of biomarkers detected by the LBS has an association with clinical outcome. Clinical outcome will be assessed for all patients (between 40 and 70 patients will be included in this study) by telephone follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nick West, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridgeshire, United Kingdom